CLINICAL TRIAL: NCT02447900
Title: Proof of Concept Study Evaluating Safety and Performance of a Gel Marker (BioXmark) Used for Image Guidance in Deep Inspiration Breathhold Radiotherapy (DIBH IGRT) in Patients With Locally Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Marker Guided Breathhold Radiotherapy in NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Steen Riisgaard Mortensen (Other)
Responsible Party: Sponsor-Investigator, Steen Riisgaard Mortensen, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 310-01
Record Dates: First submitted 2015-05-12; First posted 2015-05-19 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other)
  Interventions: Device: BioXmark

INTERVENTIONS:
Device: BioXmark

SUMMARY:
Proof of concept study evaluating safety and performance of a gel marker (BioXmark) used for image guidance in deep inspiration breathhold radiotherapy (DIBH IGRT) in patients with locally advanced non-small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion criteria

* Age > 18 years old
* Histologically confirmed non-small cell lung cancer (NSCLC)
* Stage T1-4N1-3M0
* Performance status ≤ 2
* Inoperable
* FEV1 ≥ 1 l
* Ability to hold deep inspiration breathhold for > 15 seconds
* Accepting treatment at Rigshospitalet
* Eligible for concomitant chemo-radiotherapy
* If a woman is of childbearing potential, a negative pregnancy test must be documented
* Ability to understand the given information
* Signed written consent for inclusion into the study

Exclusion criteria

* Prior thoracic radiotherapy
* Allergy to Iodine or iodine based contrast
* In the opinion of the investigator, the patient will not be able to follow the study procedures or is considered not eligible for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Visibility of the injected gel marker during the course of radiotherapy delivery | 3 months
  Stability of the geometrical configuration and visibility of the injected gel marker in 2D kV x-rays and CBCT (cone-beam computed tomography) acquired throughout the treatment course and quantified by vectors and contrast to noise ratio (CNR)
Number of pneumothoraxes in relation to placement procedure of the gel | 0-1 week after placement of gel
  Counting number of pneumothoraxes caused in relation to the placement procedure of the gel

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Denmark, Copenhagen, Denmark